CLINICAL TRIAL: NCT02997709
Title: Collection and Measurement of Blood and Imaging Biomarkers in Patients Undergoing Standard Primary and Postoperative Radiotherapy for Prostatic Neoplasms - The Miami CoMBINe Trial
Brief Title: Collection and Measurement of Biomarkers in Prostate Cancer Radiotherapy Patients
Acronym: COMBINE
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Bankhead-Coley Florida Biomedical Research Program (Unknown)
Responsible Party: Principal Investigator, Alan Pollack, MD, PhD, Professor, University of Miami
Other Study IDs: 20150452; NCI-2019-08552 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP))
Record Dates: First submitted 2016-12-15; First posted 2016-12-20 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Circulating Tumor Cells; CTCs; Androgen Deprivation Therapy; ADT
MeSH Terms: conditions — Prostatic Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected pre-RT and in post-RT follow-up for research. Plasma and serum, as well as red cells and lymphocytes (buffy coat) will be collected. The procedures will evolve with new developments, such as the ability to isolate viable CTCs for cell culture and gene expression analyses. Excess blood that is not processed for CTC or biomarkers will be stored for future research.
  Genomic studies, including genome-wide association studies (GWAS), will examine associations with health conditions are planned. Gene expression from mpMRI-defined high risk tumor regions will be related to pathologic parameters and RT response. Using a 1.4M marker oligonucleotide microarray that is essentially a whole transcriptome assay, selected pathways will be examined in pre-Tx biopsies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radiation Therapy Group: Participants with prostate cancer diagnosis who are scheduled to undergo radiotherapy (definitive or palliative) with or without the addition of Androgen Deprivation Therapy (ADT) will be evaluated
- Prostatectomy Group: Participants with prostate cancer diagnosis who are scheduled to undergo prostatectomy will be evaluated.

SUMMARY:
The purpose of this research study is to learn about: 1) How standard radiation treatment to prostate (primary radiotherapy) or the pelvis after prostatectomy (postoperative radiotherapy) may cause changes in MRI and PET imaging traits that might be used in the future to predict response. 2) Comparison of such MRI and PET imaging traits with the number of circulating tumor cells (CTCs) present in the blood prior to treatment and the changes in these counts after treatment. 3) How MRI and PET imaging characteristics and changes are related to the expression of genes in the cancer tissue obtained before treatment from prostate biopsy or a prior prostatectomy before treatment. 4) How the response of prostate cancer treatment relates to the imaging and CTC changes.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic confirmation of prostate cancer.
2. Any T-stage.
3. By imaging or clinical criteria, any patient with disease staging of N0/N1 and M0/M1.

   * Patients with metastatic disease are encouraged to participate.
4. Any Gleason Score will be eligible.
5. Androgen deprivation therapy (ADT) is at the discretion of the treating physician, but must be declared as none, short-term, long-term, or extended prior to enrollment. The length is calculated from the LHRH (agonist injection). If ADT is planned (based on treating physician preference), the following restrictions apply:

   * Short term ADT is defined as ≤ 7 months;
   * Long term ADT is defined as > 7 months and ≤ 36 months;
   * Extended ADT is defined as >36 months (e.g., M1 patients).
6. Prostate-specific antigen (PSA) ≤100 ng/mL within (+/-) 4 months of signing of consent. If PSA was above 100 and drops to <100 with antibiotics, this is acceptable for enrollment.
7. No previous pelvic radiotherapy.
8. The ability to understand and the willingness to sign a written informed consent document
9. Zubrod performance status ≤ 2 (Karnofsky or ECOG performance status may be used to estimate Zubrod):
10. Age ≥ 30 at signing of consent.
11. Subjects must be planned to receive radiation therapy or to undergo prostatectomy.
12. Subjects treated primarily with RT are recommended to have had an MUFgBx prior to radiation treatment.

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult men with a prostate cancer diagnosis.
Study Population: Adult men with a prostate cancer diagnosis undergoing standard of care treatment at the University of Miami.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2016-06-24 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of Pre- and Post-Treatment Quantitative Imaging Parameters to Changes in Circulating Tumor Cells Over Time in Study Participants. | Baseline, within 8 Days Prior to End of RT, 3 months Post-RT, 9 months and 2-2.5 Years Post-RT
  Pre-Treatment and Post-Treatment quantitative imaging parameters will be associated with circulating tumor cell (CTC) changes over time in prostate cancer (PCa) patients who receive treatment with RT ± androgen deprivation therapy (ADT) or prostatectomy per standard of care. CTC and quantitative imaging changes will be determined at each of the planned research acquisition time points (8 days prior to completion of radiation therapy (RT), 3 months post-RT, 9 months post-RT, and 2-2.5 years post-treatment) comparing to the Baseline.

SECONDARY OUTCOMES:
Relationship of CTC changes and/or quantitative imaging parameter changes to patient outcome (biochemical and clinical disease failure). | Between Baseline and 2-2.5 Years Post-RT
  CTC changes between baseline and 2-2.5 years will be compared with 2-2.5 year biopsy positivity status (positive vs. negative) for patients whose baseline and 2-2.5 year biopsy samples are available. CTC changes from two different time points will be tested for significance using t-test by 2-2.5 year biopsy positivity status. Correlation structures between CTC and imaging parameters will be analyzed using linear mixed-effect model by 2-2.5 year biopsy positivity status.
Relationship of Androgen Deprivation Therapy (ADT) status to quantitative imaging features and/or CTC levels in patients | Between Baseline and 2-2.5 Years Post-RT
  Change of CTC and imaging parameters at a specific time point from baseline will be compared by ADT status (yes vs. no) using t-test. Correlation structure between CTC and imaging parameters will be analyzed using linear mixed-effect model by ADT status.
Relationship of quantitative imaging characteristics and/or CTC changes with other tissue biomarkers obtained from the pre-treatment MRI ultrasound (US) fusion guided prostate biopsy or prostatectomy tissue in those treated primarily. | Between Baseline and 2-2.5 Years Post-RT
  Gene expression data obtained at baseline will be analyzed in order to investigate the relationship between the gene expression and the following: CTCs, mpMRI imaging parameters, histopathological tumor parameters, and biochemical/clinical failure.
  CTC changes between baseline and 2-2.5 years will be compared with 2-2.5 year biopsy positivity status (positive vs. negative) for patients whose baseline and 2-2.5 year biopsy samples are available. CTC changes from two different time points will be tested for significance using t-test by 2-2.5 year biopsy positivity status. Changes in gene expression and imaging parameters will be analyzed in the same manner. Correlation structures between CTC and imaging parameters; CTC and gene expression; and imaging parameters and gene expression will be analyzed using linear mixed-effect model by 2-2.5 year biopsy positivity status.
Comparison of changes in CTCs to endpoint prostate research biopsy status. | Between Baseline and 2-2.5 Years Post-RT
  In patients who have undergone the MRI-US fusion guided biopsy (MUFgBx) at 2-2.5 years after all planned treatment, to investigate the relationship of circulating tumor cell (CTC) changes with the endpoint of research prostate biopsy status (only for those who are treated primarily with RT, who are not on indefinite ADT and who agree to this prostate early "endpoint" biopsy).
Comparison of changes in quantitative imaging characteristics to endpoint prostate research biopsy status. | Between Baseline and 2-2.5 Years Post-RT
  In patients who have undergone the MRI-US fusion guided biopsy (MUFgBx) at 2-2.5 years after all planned treatment, to investigate the relationship of quantitative imaging characteristics with the endpoint of research prostate biopsy status (only for those who are treated primarily with RT, who are not on indefinite ADT and who agree to this prostate early "endpoint" biopsy).
Comparison of changes in gene expression patterns to endpoint prostate research biopsy status. | Between Baseline and 2-2.5 Years Post-RT
  In patients who have undergone the MRI-US fusion guided biopsy (MUFgBx) at 2-2.5 years after all planned treatment, to investigate the relationship of pretreatment biopsy tissue gene expression patterns with the research endpoint of prostate biopsy status (only for those who are treated primarily with RT, who are not on indefinite ADT and who agree to this prostate early "endpoint" biopsy).
Determination of the added value of PET/CT using newer tracers to MRI | Between Baseline and 2-2.5 Years Post-RT
  PET/CT using newer tracers (fluciclovine, prostate-specific membrane antigen (PSMA), or Choline) to MRI may add value in the above secondary analyses. The investigators hypothesize that targeted PET agents will enhance the rate of accuracy of mpMRI in establishing high risk areas in the prostate, prostate bed, and pelvic lymph nodes, as well as provide unique information on early metastatic disease.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Pollack, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No